CLINICAL TRIAL: NCT07226388
Title: Hemiarthroplasty Versus Total Shoulder Arthroplasty for the Treatment of Glenohumeral Osteoarthritis: The Impact of Modern Implant Options
Brief Title: Pyrocarbon Hemiarthroplasty Versus Total Shoulder Arthroplasty for the Treatment of Glenohumeral Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Benjamin Zmistowski, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202501233
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Glenohumeral Osteoarthritis
Keywords: hemiarthroplasty; anatomic total shoulder arthroplasty; pyrocarbon
MeSH Terms: interventions — Hemiarthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hemiarthroplasty with pyrocarbon (Active Comparator)
  Interventions: Device: Hemiarthroplasty with pyrocarbon
- Anatomic total shoulder arthroplasty (Active Comparator)
  Interventions: Device: Anatomic total shoulder arthroplasty

INTERVENTIONS:
Device: Hemiarthroplasty with pyrocarbon — Hemiarthroplasty with pyrocarbon
  Arms: Hemiarthroplasty with pyrocarbon
Device: Anatomic total shoulder arthroplasty — Anatomic total shoulder arthroplasty
  Arms: Anatomic total shoulder arthroplasty

SUMMARY:
This is a multi-center study assessing postoperative outcomes associated with hemiarthroplasty with pyrocarbon (hPYC) versus anatomic total shoulder arthroplasty (aTSA). Once eligibility criteria is met, the subject will be randomized to one of the two study arms. Subjects will be followed for ten years. Clinical and patient-reported outcome measures (PROMs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English language
2. Willing to sign an informed consent form
3. Willing to comply with all study procedures and be available for the duration of the study
4. Age 40 to 65 years
5. In good general health as evidenced by medical history
6. Surgical indication of glenohumeral osteoarthritis 7. In the opinion of the surgeon, there is clinical equipoise for the subject to be implanted with a humeral hemiarthroplasty with pyrocarbon or anatomic total shoulder arthroplasty

Exclusion Criteria:

1. Presence of Walch Type C or D glenoid
2. Presence of a glenoid that could not be reconstructed with the anatomic glenoid resurfacing components
3. Presence of extreme preoperative glenoid deformity including uniplanar retroversion deformity >30 o or severe biplanar deformity (retroversion >20 o and inclination > 10 o).
4. Workers' compensation case
5. Presence of full-thickness rotator cuff tear
6. Known allergic reactions to components of the study product(s)
7. History of consistent narcotic use within three months of surgery
8. History of chronic oral corticosteroid use
9. History or current drug or alcohol abuse
10. In the surgeon's opinion, the subject will be non-compliant with the study protocol.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2038-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Single Assessment Numeric Evaluation score | 2-years
  Assess shoulder pain and function. The score ranges from 0 to 100 with higher scores indicating a better shoulder function and less pain.

SECONDARY OUTCOMES:
American Shoulder and Elbow Visual Analog Pain Score | 2-weeks, 3-months, 6-months, 1-year, 2-years, 5-years, 10-years
  Assess pain relief. Range: 0-10. Zero is equivalent to no pain and 10 indicates the worst possible pain
Forgotten Joint score | 2-weeks, 3-months, 6-months, 1-year, 2-years, 5-years, 10-years
  Assess shoulder function. The total score ranges from 0 to 100 with higher scores indicating a high degree of forgetting the artificial joint.
Range of motion | 2-weeks, 3-months, 6-months, 1-year, 2-years, 5-years, 10-years
  Assess shoulder motion. Subjects will have their shoulder range of motion measured in degrees.
Assess rates of glenoid erosion | 2-years, 5-years, 10-years
  Assess rates of glenoid erosion associated with pyrocarbon hemiarthroplasty
Assess rates of aseptic glenoid loosening | 2-years, 5-years, 10-years
  Assess rates of aseptic glenoid loosening associated with anatomic total shoulder arthroplasty
Single Assessment Numeric Evaluation Score | 5-years, 10-years
  Assess shoulder pain and function. The score ranges from 0 to 100 with higher scores indicating a better shoulder function and less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Zmistowski, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States